CLINICAL TRIAL: NCT05154409
Title: Blood and Urine Sample Collection From Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Evotec International GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: EVT_CTC_01
Record Dates: First submitted 2021-07-13; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to obtain blood and urine samples from healthy volunteers to serve as a healthy control group for cross-cohort comparisons.

DETAILED DESCRIPTION:
The aim of the study is to obtain peripheral venous blood samples and a urine sample from 100 healthy volunteers on one day at three different times of the day, to serve as a healthy control group for cross-cohort comparisons.

With the help of the urine and blood samples obtained in this context, a cohort of a healthy collective is to be established for further research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 40-70 years.
* Caucasian
* Non-smokers or ex-smokers
* Body Mass Index (BMI): ≥18.5 and ≤32 kg/m2
* Presence of a negative SARS-CoV-2 PCR test.

Exclusion Criteria:

* Complaints that may indicate the presence of an infection, including Covid-19.
* Pathological alcohol consumption.
* Positive alcohol breath test at the preliminary examination.
* Alcohol consumption within the last 24 hours before the start of sampling.
* History of drug dependence.
* Positive urine drug test during the preliminary examination.
* Clinically significant acute or chronic disease. In particular, chronic inflammation, rheumatological and other autoimmune diseases, diabetes and other metabolic diseases.
* Indications in the medical history or during the medical examination that may jeopardize the safety of the study participant by participating in the study.
* History of relevant clinically significant cardiovascular disorders or clinically relevant hyper- or hypotension or clinically relevant brady- or tachycardia at screening as assessed by an investigator.
* Heart rate <45/min after 5 minutes in a quiet sitting position.
* Heart rate >100/min after 5 minutes in a quiet sitting position.
* Systolic blood pressure of > 170 mmHg or < 90 mmHg.
* Diastolic blood pressure of > 95 mmHg and/or < 60 mmHg.
* Regular use of prescription medication within 3 months prior to inclusion in the research project.
* Use of non-prescription medications within 3 days prior to inclusion in the research project.
* Presence of clinically significant food intolerance and/or food allergy as assessed by the investigator.
* Medically relevant previous operations.
* Condition following radio- or chemotherapy.
* History of oncological diseases.
* Blood and/or plasma donation within the last 30 days prior to sample collection.
* Pregnant or nursing female.
* Employees of study site.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers who met all inclusion and none of the exlusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Collection of blood samples from healthy volunteers to serve as a healthy control group. | 1 day
  There are no primary endpoints planned; endpoints will be specified in the individual research projects that will utilize the blood samples as a control group.
Collection of urine samples from healthy volunteers to serve as a healthy control group. | 1 day
  There are no primary endpoints planned; endpoints will be specified in the individual research projects that will utilize the urine samples as a control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Peradziryi, Study Chair — Hanna.Peradziryi@evotec.com
Locations (1):
- CTC North, Hamburg, Germany